CLINICAL TRIAL: NCT01245556
Title: A Phase 1 Study of a RAF Inhibitor (BMS-908662) Administered in Combination With Immunotherapy (Ipilimumab) in Subjects With Unresectable Stage III or Stage IV Melanoma
Brief Title: Safety and Efficacy Study of BMS-908662 in Combination With Ipilimumab in Subjects With Advanced Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA206-005
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — BMS 908662; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BMS-908662 or Ipilimumab (A) (Experimental)
  Interventions: Drug: BMS-908662; Drug: Ipilimumab
- BMS-908662 or Ipilimumab (B) (Experimental)
  Interventions: Drug: BMS-908662; Drug: Ipilimumab

INTERVENTIONS:
Drug: BMS-908662 — Capsules, Oral, escalating doses starting at 25 mg, Q 12 h daily, Continuously
  Arms: BMS-908662 or Ipilimumab (A)
Drug: BMS-908662 — Capsules, Oral, escalating doses starting at 25 mg Q 12 h daily for 3 weeks with 3 weeks interval for 4 cycles, then Q12 h daily for 3 weeks every 12 weeks, Continuously
  Arms: BMS-908662 or Ipilimumab (B)
Drug: Ipilimumab — Vial, IV, escalating doses starting at 3 mg/kg, Once every 3 weeks for 6 weeks, then once every 12 weeks, Continuously
  Arms: BMS-908662 or Ipilimumab (A)
Drug: Ipilimumab — Vial, IV, escalating doses starting at 3 mg/kg, Once every 6 weeks for 4 cycles, then once every 12 weeks, Continuously
  Arms: BMS-908662 or Ipilimumab (B)

SUMMARY:
The purpose of the study is to identify a safe and tolerable dose of BMS-908662 in combination with ipilimumab; and then to evaluate the anti-tumor response to BMS-908662 when administered in combination with ipilimumab.

ELIGIBILITY:
Inclusion:

* Male and female subjects ≥ 18 years of age with a histologic or cytologic diagnosis of Stage III or Stage IV (unresectable) melanoma
* Enrollment to cohort expansion will be limited to only those subjects whose tumors demonstrate the B-Raf V600E mutation
* ECOG ≤ 1
* Adequate organ & marrow function

Exclusion:

* Uncontrolled or significant cardiovascular disease
* Cohort expansion: Prior therapy with a RAF inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Toxicity will be evaluated according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE) version 3 | Assessments approximately every 3 weeks throughout the duration of the trial

SECONDARY OUTCOMES:
Efficacy as determined by estimates of objective response rates and response duration | Efficacy measured every 6 weeks until week 48, then every 12 weeks
PK for BMS-908662 as determined by minimum and maximum observed concentrations, time of maximum observed concentration, area under the concentration curve for one dosing interval and the accumulation index | PK measured during first 4 weeks on study
PD will be assessed by evaluating markers of RAS/RAF pathway activity | PD assessed during the first 4 weeks on study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Jedd D. Wolchok, Md,Phd, New York, New York

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx